CLINICAL TRIAL: NCT01063881
Title: The Asia-Pacific Flexible Dose Study of Dapoxetine and Patient Satisfaction in Premature Ejaculation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016561; R096769PRE3009 (Other: Johnson & Johnson Pte Ltd); PASSION (Other: Johnson & Johnson Pte Ltd)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Sexual Dysfunction, Physiological
Keywords: Sexual Dysfunction, physiological; R096769; Dapoxetine; Phase 3b; Premature Ejaculation
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Premature Ejaculation | interventions — dapoxetine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No

ARMS (1):
- Dapoxetine (Experimental): Starting dose is one 30-mg tablet taken approximately 1-3 hours prior to sexual activity may be increased after 4 weeks to 60mg taken for 12 weeks. The maximum recommended dosing frequency is once every 24 hours.
  Interventions: Drug: Dapoxetine

INTERVENTIONS:
Drug: Dapoxetine — Starting dose is one 30-mg tablet taken approximately 1-3 hours prior to sexual activity, may be increased after 4 weeks to 60mg, taken for 12 weeks. The maximum recommended dosing frequency is once every 24 hours.

SUMMARY:
The purpose of the study is to measure the efficacy of flexible dosing of dapoxetine in a setting similar to routine clinical practice.

DETAILED DESCRIPTION:
This is a prospective, interventional study to evaluate efficacy and safety of flexible dose dapoxetine as Premature Ejaculation (PE) Therapy. The total study duration will be 16 weeks, composed of a 2-week pretreatment phase and a 12-week open-label treatment phase, followed by a telephone contact two weeks after Week 12 to follow-up adverse events. At Visit 1 (Screening) standardized assessment tool or patient questionnaires will be used to determine which of those patients with erectile dysfunction/premature ejaculation are eligible to participate in this study. Once enrolled the patient and his partner are expected to attempt sexual intercourse a minimum of 2 times (at least 24 hours apart) and to complete a Baseline Event Log. Starting at Visit 2 (Baseline), the patient (and partner) will complete the Premature Ejaculation Profile (PEP) at the beginning of every treatment visit for the duration of the study. Patients will be started on study drug instructed to take 1 tablet of dapoxetine 30 mg, as needed, 1 to 3 hours prior to sexual activity. The need for adjustments in the dose of dapoxetine, as well as to assess the occurrence of adverse events and concomitant therapy use will be assessed approximately every 4 weeks. Patients will complete Treatment Event Logs during each dosing throughout the open-label treatment phase. Patients who have their dose increased to 60 mg, will be scheduled for a telephone consultation 1 week after to determine how the dose change is tolerated. At Visit 5 (Final Visit/Week 12/Early Termination), the patients and partners will complete several standardized assessment questionnaires have all final visit procedures performed and schedule a telephone follow up contact to evaluate any adverse events. The starting dose of dapoxetine is 30 mg (one 30-mg tablet), taken approximately 1 to 3 hours prior to sexual activity. The dose may be increased after 4 weeks to 60 mg taken. The maximum recommended dosing frequency is once every 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be heterosexual males and in a stable monogamous, sexual relationship with a female partner for at least 6 months
* must score =11 in the Premature Ejaculation Diagnostic Tool (PEDT)
* Must have a self-estimated intravaginal ejaculatory latency time (IELT) of = 2 minutes
* Must have an International Index of Erectile Dysfunction (IIEF) score a total of > or = to 21 in 6 questions from the IIEF used to assess for the absence of moderate to severe erectile dysfunction (ED)
* Premature ejaculation is not exclusively due to the direct effects of a substance (e.g., withdrawal from opioids)
* Must be in good general health with no clinically significant abnormalities as determined by medical history, physical examination, and clinical lab results
* Must have a blood pressure =180 mmHg systolic and =100 mmHg diastolic at screening and at the baseline visit
* Patient's partner must not be pregnant at screening as pregnancy might affect sexual activity
* Participants and partners must agree to attempt sexual intercourse at least 2 times (with a minimum of 24 hours between each event) during the 2-week baseline period and at least 4 times per month during the remainder of the study.

Exclusion Criteria:

* History of or current major psychiatric disorder such as mood disorder, anxiety disorder, schizophrenia, mania, suicidal ideation, other psychotic disorder
* History of alcohol abuse and dependence, non-alcohol psychoactive substance use disorder (except for caffeine or nicotine/tobacco)
* Suspected history of illicit or recreational drug use
* Known history of moderate to severe renal impairment

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2010-05-22 (Actual); Primary Completion 2011-06-14 (Actual); Study Completion 2011-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (13):
- Australia (3):
  - Malvern
  - St Leonards
  - Sydney
- South Korea (8):
  - Busan
  - Daegu
  - Gwangju
  - Incheon
  - Jeonju
  - Jinju
  - Seoul
  - Wŏnju
- Thailand (2):
  - Bangkok
  - Chiang Mai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 285 patients were enrolled in the study, of which 281 patients received at least 1 dose of study drug were included in the safety analysis set (Dapoxetine 30 mg only [144 patients], Dapoxetine 30 t0 60 mg [124 patients] and Dapoxetine 30 to 60 to 30 mg [13 patients]).
Groups:
- Dapoxetine 30 mg Only: Patients who took dapoxetine 30 mg throughout the study. The maximum recommended dosing frequency is once every 24 hours. The duration of the treatment period was 12 weeks.
- Dapoxetine 30 to 60 mg: Patients who started on dapoxetine 30 mg and required an increase to dapoxetine 60 mg for the remainder of the study. The maximum recommended dosing frequency is once every 24 hours. The duration of the treatment period was 12 weeks.
- Dapoxetine 30 to 60 to 30 mg: Patients who started on dapoxetine 30 mg, required an increase to dapoxetine 60 mg but later required a down-titration (decrease) to dapoxetine 30 mg for the remainder of the study. The maximum recommended dosing frequency is once every 24 hours. The duration of the treatment period was 12 weeks.
Period: Overall Study
Arm/Group | Dapoxetine 30 mg Only | Dapoxetine 30 to 60 mg | Dapoxetine 30 to 60 to 30 mg
Started | 147 | 125 | 13
Completed | 92 | 114 | 12
Not Completed | 55 | 11 | 1
Not completed — Adverse Event | 12 | 2 | 0
Not completed — Lost to Follow-up | 13 | 7 | 1
Not completed — Withdrawal by Subject | 25 | 1 | 0
Not completed — Reason for not completed not specified | 5 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dapoxetine 30 mg Only: 144 of 147 patients took at least 1 dose of dapoxetine 30 mg throughout the study. The maximum recommended dosing frequency is once every 24 hours. The duration of the treatment period was 12 weeks.
- Dapoxetine 30 to 60 mg: 124 of 125 patients took at least one dose of dapoxetine 30 mg and required an increase to dapoxetine 60 mg for the remainder of the study. The maximum recommended dosing frequency is once every 24 hours. The duration of the treatment period was 12 weeks.
- Dapoxetine 30 to 60 to 30 mg: 13 patients took at least one dose of dapoxetine 30 mg, required an increase to dapoxetine 60 mg but later required a down-titration (decrease) to dapoxetine 30 mg for the remainder of the study. The maximum recommended dosing frequency is once every 24 hours. The duration of the treatment period was 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Dapoxetine 30 mg Only | Dapoxetine 30 to 60 mg | Dapoxetine 30 to 60 to 30 mg | Total
Number analyzed (Participants) | 144 | 124 | 13 | 281
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 142 | 121 | 13 | 276
  >=65 years | 2 | 3 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (10.43) | 46.9 (10.47) | 41.1 (7.77) | 45.9 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 144 | 124 | 13 | 281
Baseline BMI [Mean (Standard Deviation); unit: kg/cm^2] | 24.7 (2.79) | 25.3 (3.20) | 23.9 (2.78) | 24.9 (2.99)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Described Their Premature Ejaculation (PE) as At Least "Slightly Better" in Response to Dapoxetine Treatment
Description: The "Clinical Global Impression of Change" (CGIC), a patient-reported scale was used to assess the patient's improvement with premature ejaculation (PE) since initiating treatment with dapoxetine. Patients were asked: "Compared to the start of the study, would you describe your premature ejaculation (PE) problem as: Much worse, Worse, Slightly worse, No change, Slightly better, Better, or Much better?" The number of patients who described improvement with their PE of at least "slightly better" after 12 weeks of treatment with dapoxetine are provided in the table below.
Time Frame: Week 12
Population: The full analysis set (FAS) included all patients who took at least one dose of study drug and completed at least one assessment of efficacy.
Measure: Number; unit: Patients
Groups:
- Dapoxetine (Week 12): Patients took Dapoxetine at a starting dose of one 30-mg tablet approximately 1-3 hours prior to sexual activity. After 4 weeks of treatment, the dosage of dapoxetine may have been increased to 60mg. The maximum recommended dosing frequency is once every 24 hours. The total duration of treatment was 12 weeks.
Arm/Group | Dapoxetine (Week 12)
Number analyzed (Participants) | 257
Patients | 228

2. Secondary Outcome: The Patient's Level of Control Over Ejaculation
Description: The Premature Ejaculation Profile (PEP), a patient-reported outcome measure was used to rate the patient's level of control over intercourse on a 5-point scale. Patients were asked: "Over the past month, was your level of control over ejaculation Very poor, Poor, Fair, Good, or Very Good?" The number of patients who rated their level of control over ejaculation before treatment and after 12 weeks of treatment with dapoxetine are provided in the table below.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: Patients
Groups:
- Dapoxetine (Baseline): Baseline measures were taken before administration of treatment.
Arm/Group | Dapoxetine (Baseline) | Dapoxetine (Week 12)
Number analyzed (Participants) | 274 | 278
Patients
  Very poor | 120 | 22
  Poor | 132 | 57
  Fair | 20 | 77
  Good | 2 | 101
  Very good | 0 | 21

3. Secondary Outcome: The Patient's Level of Satisfaction With Intercourse
Description: The Premature Ejaculation Profile (PEP), a patient-reported outcome measure was used to rate the patient's level of satisfaction with intercourse on a 5-point scale. Patients were asked: "Over the past month, was your satisfaction with sexual intercourse Very poor, Poor, Fair, Good, or Very Good?" The number of patients who rated their level of satisfaction with control over ejaculation at before treatment and after 12 weeks of treatment with dapoxetine are provided in the table below.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Dapoxetine (Baseline) | Dapoxetine (Week 12)
Number analyzed (Participants) | 274 | 278
Patients
  Very poor | 63 | 14
  Poor | 152 | 40
  Fair | 53 | 89
  Good | 6 | 105
  Very good | 0 | 30

4. Secondary Outcome: The Patient's Level of Personal Distress Related to the Speed of Ejaculation
Description: The Premature Ejaculation Profile (PEP), a patient-reported outcome measure was used to rate the patient's level of distress related to the speed of ejaculation. Patient's were asked: "Over the past month, how distressed were you by how fast you ejaculated during sexual intercourse? Not at all, A little bit, Moderately, Quite a bit, Extremely." The number of patients who rated their level of personal distress related to the speed of ejaculation before treatment and after 12 weeks of treatment with dapoxetine are provided in the table below.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Dapoxetine (Baseline) | Dapoxetine (Week 12)
Number analyzed (Participants) | 274 | 278
Patients
  Not at all | 2 | 66
  A little bit | 32 | 89
  Moderately | 32 | 66
  Quite a bit | 140 | 40
  Extremely | 68 | 17

5. Secondary Outcome: The Patient's Degree of Interpersonal Difficulty Related to the Speed of Ejaculation
Description: The Premature Ejaculation Profile (PEP), a patient-reported outcome measure was used to rate the patient's level of interpersonal difficulty related to the speed of ejaculation. Patient's were asked: "Over the past month, to what extent did how fast you/your partner ejaculated during sexual intercourse cause difficulty in your relationship with your partner? Not at all, A little bit, Moderately, Quite a bit, or Extremely?" The number of patients who rated their level of interpersonal difficulty before treatment and after 12 weeks of treatment with dapoxetine are provided in the table below.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Dapoxetine (Baseline) | Dapoxetine (Week 12)
Number analyzed (Participants) | 274 | 278
Patients
  Not at all | 12 | 87
  A little bit | 40 | 82
  Moderately | 78 | 65
  Quite a bit | 113 | 37
  Extremely | 31 | 7

6. Secondary Outcome: Patient Responses to Improvement With Their Premature Ejaculation After 12 Weeks of Treatment With Dapoxetine
Description: The "Clinical Global Impression of Change" (CGIC), a patient-reported scale was used to assess the patient's improvement with premature ejaculation (PE) since initiating treatment with dapoxetine. Patients were asked: "Compared to the start of the study, would you describe your premature ejaculation (PE) problem as: Much worse, Worse, Slightly worse, No change, Slightly better, Better, or Much better?" The number of patients reporting improvement in their PE by category of the CGIC scale after 12 weeks of treatment with dapoxetine are provided in the table below.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Dapoxetine (Week 12)
Number analyzed (Participants) | 257
Patients
  Much worse | 0
  Worse | 0
  Slightly worse | 4
  No change | 25
  Slightly better | 94
  Better | 101
  Much better | 33

7. Secondary Outcome: The Number of Patients Who Described Their Premature Ejaculation (PE) as At Least "Slightly Better" in Response to Dapoxetine Treatment (Subgroups by Dosage)
Description: The "Clinical Global Impression of Change" (CGIC) was used to assess the patient's improvement with premature ejaculation (PE) since initiating treatment with dapoxetine. The data provided below represent the number of patients who reported at least a slightly better response to treatment by the dose of dapoxetine they received in the study. This was a single-arm, open-label, non-randomized study in which "subgroup by dosage" was categorized based on dose-titration patterns observed during the course of the treatment period.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Dapoxetine 30 mg Only | Dapoxetine 30 to 60 mg | Dapoxetine 30 to 60 to 30 mg
Number analyzed (Participants) | 141 | 124 | 13
Patients | 109 | 107 | 12

8. Secondary Outcome: The Number of Patients Who Described Their Premature Ejaculation (PE) as At Least "Slightly Better" in Response to Dapoxetine Treatment (Subgroups by Disease Type)
Description: The "Clinical Global Impression of Change" (CGIC) was used to assess the patient's improvement with premature ejaculation (PE) since initiating treatment with dapoxetine. The data provided below represent the number of patients who reported at least a "slightly better" response to treatment when grouped by type of PE disease (patients with life-long PE and patients with acquired PE). This was a single-arm, open-label, non-randomized study where patients were categorized based their PE disease after enrollment in the study.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Patients
Groups:
- Dapoxetine (Patients With Life-long PE, Week 12); Dapoxetine (Patients With Acquired PE, Week 12): Patients took Dapoxetine at a starting dose of one 30-mg tablet approximately 1-3 hours prior to sexual activity. After 4 weeks of treatment, the dosage of dapoxetine may have been increased to 60mg. The maximum recommended dosing frequency is once every 24 hours. The total duration of treatment was 12 weeks.
Arm/Group | Dapoxetine (Patients With Life-long PE, Week 12) | Dapoxetine (Patients With Acquired PE, Week 12)
Number analyzed (Participants) | 115 | 163
Patients | 95 | 133

9. Secondary Outcome: The Number of Patients Who Described Their Premature Ejaculation (PE) as At Least "Slightly Better" in Response to Dapoxetine Treatment (Subgroups by Intravaginal Ejaculation Latency Time [IELT])
Description: The "Clinical Global Impression of Change" (CGIC) was used to assess the patient's improvement with premature ejaculation (PE) since initiating treatment with dapoxetine. The data provided below represent the number of patients who reported at least a "slightly better" response to treatment when grouped by intravaginal ejaculation latency time (patients with an IELT of < 1 minute and patients with an IELT of > 1 minute). This was a single-arm, open-label, non-randomized study where patients were categorized based on IELT after enrollment in the study.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Patients
Groups:
- Dapoxetine (Patients With IELT <1 Minute, Week 12); Dapoxetine (Patients With IELT >1 Minute, Week 12): Patients took Dapoxetine at a starting dose of one 30-mg tablet approximately 1-3 hours prior to sexual activity. After 4 weeks of treatment, the dosage of dapoxetine may have been increased to 60mg. The maximum recommended dosing frequency is once every 24 hours. The total duration of treatment was 12 weeks.
Arm/Group | Dapoxetine (Patients With IELT <1 Minute, Week 12) | Dapoxetine (Patients With IELT >1 Minute, Week 12)
Number analyzed (Participants) | 138 | 140
Patients | 110 | 118

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the duration of the study.
Groups:
- Depoxetine (DPX) 30 mg Only: Patients who took dapoxetine 30 mg throughout the study. The maximum recommended dosing frequency is once every 24 hours. The duration of the treatment period was 12 weeks.
- Depoxetine (DPX) 30 to 60 mg: Patients who started on dapoxetine 30 mg and required an increase to dapoxetine 60 mg for the remainder of the study. The maximum recommended dosing frequency is once every 24 hours. The duration of the treatment period was 12 weeks.
- Depoxetine (DPX) 30 to 60 to 30 mg: Patients who started on dapoxetine 30 mg, required an increase to dapoxetine 60 mg but later required a down-titration (decrease) to dapoxetine 30 mg for the remainder of the study. The maximum recommended dosing frequency is once every 24 hours. The duration of the treatment period was 12 weeks.
Arm/Group | Depoxetine (DPX) 30 mg Only | Depoxetine (DPX) 30 to 60 mg | Depoxetine (DPX) 30 to 60 to 30 mg
Serious Adverse Events (participants affected / at risk) | 2/144 | 0/124 | 0/13
Other Adverse Events (participants affected / at risk) | 62/144 | 57/124 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Depoxetine (DPX) 30 mg Only (N=144) | Depoxetine (DPX) 30 to 60 mg (N=124) | Depoxetine (DPX) 30 to 60 to 30 mg (N=13)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Depoxetine (DPX) 30 mg Only (N=144) | Depoxetine (DPX) 30 to 60 mg (N=124) | Depoxetine (DPX) 30 to 60 to 30 mg (N=13)
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 4 | 3 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Dry Eye (Eye disorders) | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 3 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 1
Dry Mouth (Gastrointestinal disorders) | 3 | 4 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 14 | 18 | 6
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chest Discomfort (General disorders) | 1 | 1 | 0
Chest Pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 3 | 0
Feeling Abnormal (General disorders) | 1 | 0 | 1
Local Swelling (General disorders) | 0 | 1 | 0
Sensation of Foreign Body (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Chronic Sinusitis (Infections and infestations) | 0 | 1 | 0
Ear Infection Fungal (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Latent Syphilis (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Otitis Media (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 3 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 3 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1 | 0
Blood Pressure Increased (Investigations) | 1 | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 0
Burning Sensation (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 13 | 13 | 6
Headache (Nervous system disorders) | 13 | 12 | 1
Mental Impairment (Nervous system disorders) | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 5 | 4 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Dissociation (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0
Libido Decreased (Psychiatric disorders) | 1 | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 2 | 0 | 0
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Wrinkling (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 1 | 0
Hot Flush (Vascular disorders) | 3 | 1 | 0

LIMITATIONS AND CAVEATS:
"Subgroup by dosage" was categorized based on dose-titration patterns observed during the course of the treatment period. Patients were not randomized to treatment by dosage group, disease type, or Intravaginal Ejaculation Latency Time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days